CLINICAL TRIAL: NCT03183999
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial for Evaluation of Sperm Motility Improvement Effect of Fermented Ginseng(GINST)
Brief Title: Effect of Fermented Ginseng (GINST) on Sperm Motility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jae Hoon Lee (Other)
Collaborators: Ilwha Co.,Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Jae Hoon Lee, Clinical Fellow, Severance Hospital
Organization: Severance Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2016-0288
Record Dates: First submitted 2017-05-17; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Asthenozoospermia
MeSH Terms: conditions — Asthenozoospermia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial for evaluation of sperm motility improvement effect of fermented ginseng
Who Masked: Participant, Care Provider
Masking Description: 1. Participant masking:
     To intervention arm, capsules including 160mg of fermented ginseng(GINST) ingredients will be provided. To control arm, capsules of the same shape and weight as GINST capsules will be provided. These apsules are made of a cellulose component.
  2. Care provider masking The care providers will be unaware which participant belonged to the experimental group or control group during stuty period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GINST group (Experimental): Experimental group was randomly assigned among the volunteers who met the inclusion criteria: men between the ages of 18 and 60 who had sperm motility of less than 32%. Fermented ginseng (GINST) was supplied.
  Interventions: Dietary Supplement: fermented ginseng (GINST)
- Control group (Placebo Comparator): Control group was randomly assigned among the volunteers who met the inclusion criteria: men between the ages of 18 and 60 who had sperm motility of less than 32%. Placebo was supplied.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fermented ginseng (GINST) — Intervention group should take fermented ginseng (GINST) capsule 3 times a day, 2 capsules at one time for 12 weeks
  Arms: GINST group
Dietary Supplement: Placebo — Control group should take placebo capsule 3 times a day, 2 capsules at one time for 12 weeks
  Arms: Control group

SUMMARY:
This randomized, double-blind, placebo-controlled study aimed to evaluate the effect of ginseng(GINST) supplementation for 12 weeks on sperm motility.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled clinical trial was aimed to evaluate of sperm motility improvement effect of fermented ginseng(GINST). Experimental arm and control arm were randomly assigned among the volunteers who met the inclusion criteria: men between the ages of 18 and 60 who had sperm motility of less than 32%.

To experimental arm, capsules including 160mg of fermented ginseng(GINST) ingredients will be provided for 12 weeks. To control arm, capsules of the same shape and weight as GINST capsules will be provided. These capsules are made of a cellulose component.

Primary outcome is sperm motility. Secondary outcome are <Brief Male Sexual Function Inventory> , <Fatigue Severity Scale>, and <the Short Form (36) Health Survey> measured at baseline and end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 60 years old
* Men who have agreed to participate in this trial before the start of the study and who have written an informed consent

Exclusion Criteria:

* Those who are diagnosed and treated for hypertension (systolic blood pressure> 140mmHg and diastolic blood pressure> 90mmHg)
* Patients with a history of chemotherapy for malignant tumors
* Patients with a history of taking testosterone or antiandrogens within 1 month
* BMI> 30 or BMI <18
* Those who have the following results in the blood test: AST(aspartate aminotransferase ), ALT(Alanine transaminase) > 2 times the upper limit of reference range; Serum Creatinine> 2.0 mg / dl
* Those who ingested drugs (eg, folic acid, L-carn, HCG(human chorionic gonadotropin ), FSH(Follicle-stimulating hormone), Clomiphene, etc.) that have an effect on sperm motility within 2 weeks before the screening day.
* Persons who have received antipsychotic medication within 2 months before the screening test
* Those who have history of alcoholism or substance abuse

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Because this trial is aimed to evaluate of effect of femented ginseng on sperm motility, participant eligibility is based on biological gender.
Enrollment: 60 (Estimated)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Sperm motility | Change from baseline sperm motility at 12 weeks
  Sperm motility is evaluated by Computer-Aided Semen Analysis, or CASA. Sperm motility will be expressed as '% motile' , the percent of cells that are motile. According to WHO definition, asthenozoospermia is regarded as falling below 40% motility in this study.

SECONDARY OUTCOMES:
Quality of life | Change from baseline quality of life at 12 weeks
  Quality of life was evaluated by The Short Form (36) Health Survey(SF-36 questionnaire) at baseline and 12weeks after intervention
Fatigue questionnaire | Change from baseline Fatigue Severity Scale at 12 weeks
  Fatigue was evaluated by Fatigue Severity Scale at baseline and 12weeks after intervention
Sexual function | Change from baseline Sexual Function Inventory (questionnaire) at 12 weeks
  Sexual function was evaluated by Brief Male Sexual Function Inventory (questionnaire) at baseline and 12weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Young Sik Choi, M.D., Ph.D., Study Director — Severance Hospital, Yonsei University
Locations (3):
- South Korea (3):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwondo
  - Gil Hospital, Incheon
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen JC, Xu MX, Chen LD, Chen YN, Chiu TH. Effect of panax notoginseng extracts on inferior sperm motility in vitro. Am J Chin Med. 1999;27(1):123-8. doi: 10.1142/S0192415X9900015X. PMID 10354824
- [Background] Chen JC, Chen LD, Tsauer W, Tsai CC, Chen BC, Chen YJ. Effects of Ginsenoside Rb2 and Rc on inferior human sperm motility in vitro. Am J Chin Med. 2001;29(1):155-60. doi: 10.1142/S0192415X01000174. PMID 11321473
- [Background] Chen X, Lee TJ. Ginsenosides-induced nitric oxide-mediated relaxation of the rabbit corpus cavernosum. Br J Pharmacol. 1995 May;115(1):15-8. doi: 10.1111/j.1476-5381.1995.tb16313.x. PMID 7647970